CLINICAL TRIAL: NCT05986292
Title: A Master Protocol for Randomized, Placebo-Controlled, Phase 2 Clinical Trials of Multiple Interventions for the Treatment of Chronic Pain
Brief Title: A Master Protocol Study (LY900028) of Multiple Intervention-Specific-Appendices (ISAs) in Participants With Chronic Pain
Acronym: CPMP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 17511; H0P-MC-CPMP (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis, Knee; Diabetic Neuropathic Pain; Chronic Low-back Pain
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- LY3016859 Osteoarthritis ISA (Experimental): Participants are randomized to receive either active LY3016859 or matching placebo
  Interventions: Drug: LY3016859 ISA; Drug: Placebo
- LY3016859 Diabetic Neuropathic Pain ISA (Experimental): Participants are randomized to receive either active LY3016859 or matching placebo
  Interventions: Drug: LY3016859 ISA; Drug: Placebo
- LY3016859 Chronic Back Pain ISA (Experimental): Participants are randomized to receive either active LY3016859 or matching placebo
  Interventions: Drug: LY3016859 ISA; Drug: Placebo
- LY3556050 Osteoarthritis ISA (Experimental): Participants are randomized to receive either active LY3556050 or matching placebo
  Interventions: Drug: LY3556050 ISA; Drug: Placebo Oral
- LY3556050 Diabetic Neuropathic Pain ISA (Experimental): Participants are randomized to receive either active LY3556050 or matching placebo
  Interventions: Drug: LY3556050 ISA; Drug: Placebo Oral
- LY3556050 Chronic Back Pain ISA (Experimental): Participants are randomized to receive either active LY3556050 or matching placebo
  Interventions: Drug: LY3556050 ISA; Drug: Placebo Oral
- LY3526318 Osteoarthritis ISA (Experimental): Participants are randomized to receive either active LY3526318 or matching placebo
  Interventions: Drug: LY3526318 ISA; Drug: Placebo Oral
- LY3526318 Diabetic Neuropathic Pain ISA (Experimental): Participants are randomized to receive either active LY3526318 or matching placebo
  Interventions: Drug: LY3526318 ISA; Drug: Placebo Oral
- LY3526318 Chronic Back Pain ISA (Experimental): Participants are randomized to receive either active LY3526318 or matching placebo
  Interventions: Drug: LY3526318 ISA; Drug: Placebo Oral
- LY3857210 Osteoarthritis ISA (Experimental): Participants are randomized to receive either active LY3857210 or matching placebo
  Interventions: Drug: LY3857210 ISA; Drug: Placebo Oral
- LY3857210 Diabetic Neuropathic Pain ISA (Experimental): Participants are randomized to receive either active LY3857210 or matching placebo
  Interventions: Drug: LY3857210 ISA; Drug: Placebo Oral
- LY3857210 Chronic Back Pain ISA (Experimental): Participants are randomized to receive either active LY3857210 or matching placebo
  Interventions: Drug: LY3857210 ISA; Drug: Placebo Oral

INTERVENTIONS:
Drug: LY3016859 ISA — Administered intravenously (IV)
  Arms: LY3016859 Chronic Back Pain ISA; LY3016859 Diabetic Neuropathic Pain ISA; LY3016859 Osteoarthritis ISA
Drug: LY3556050 ISA — Administered orally
  Arms: LY3556050 Chronic Back Pain ISA; LY3556050 Diabetic Neuropathic Pain ISA; LY3556050 Osteoarthritis ISA
Drug: LY3526318 ISA — Administered orally
  Arms: LY3526318 Chronic Back Pain ISA; LY3526318 Diabetic Neuropathic Pain ISA; LY3526318 Osteoarthritis ISA
Drug: LY3857210 ISA — Administered orally
  Arms: LY3857210 Chronic Back Pain ISA; LY3857210 Diabetic Neuropathic Pain ISA; LY3857210 Osteoarthritis ISA
Drug: Placebo Oral — Placebo administered orally
  Arms: LY3526318 Chronic Back Pain ISA; LY3526318 Diabetic Neuropathic Pain ISA; LY3526318 Osteoarthritis ISA; LY3556050 Chronic Back Pain ISA; LY3556050 Diabetic Neuropathic Pain ISA; LY3556050 Osteoarthritis ISA; LY3857210 Chronic Back Pain ISA; LY3857210 Diabetic Neuropathic Pain ISA; LY3857210 Osteoarthritis ISA
Drug: Placebo — Placebo administered IV
  Arms: LY3016859 Chronic Back Pain ISA; LY3016859 Diabetic Neuropathic Pain ISA; LY3016859 Osteoarthritis ISA

SUMMARY:
The purpose of the chronic pain master protocol is to compare independent pain interventions and establish an overarching structure for the disease-state addenda (DSA) and intervention-specific appendices (ISAs). The ISAs may start independently of other ISAs as interventions become available for clinical testing.

DETAILED DESCRIPTION:
The chronic pain master protocol (CPMP) establishes entry criteria and includes DSA for osteoarthritis of the knee, chronic low back pain, and diabetic peripheral neuropathic pain. The DSA have specific study elements to appropriately define the target population and unique scales for assessment. Also, the master protocol governs ISAs that may start independently of other ISAs as interventions become available for clinical testing.

Note: Results for all outcomes are posted in the intervention records. No need for duplication.

ELIGIBILITY:
Inclusion Criteria:

* have a visual analog scale (VAS) pain value >40 and <95 at screening and prerandomization screening.
* have a history of daily pain for at least 12 weeks based on participant report or medical history
* have a value of ≤30 on the pain catastrophizing scale
* have a body mass index <40 kilogram/square meter (kg/m²) (inclusive)
* are willing to maintain a consistent regimen of any ongoing nonpharmacologic pain-relieving therapies (for example, physical therapy) and will not start any new nonpharmacologic pain-relieving therapies during study participation.
* are willing to discontinue all medications taken for chronic pain conditions, except rescue medication for the duration of the study

Exclusion Criteria:

* have second- or third-degree atrioventricular (AV) heart block or AV dissociation or history of ventricular tachycardia
* have had a procedure within the past 6 months intended to produce permanent sensory loss in the target area of interest (for example, ablation techniques)
* have surgery planned during the study for any reason, related or not to the disease state under evaluation.
* have, in the judgment of the investigator, an acute, serious, or unstable medical condition or a history or presence of any other medical illness that would preclude study participation.
* have had cancer within 2 years of baseline, except for cutaneous basal cell or squamous cell carcinoma resolved by excision.
* have fibromyalgia
* have substance use disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders (5th edition; DSM-5; American Psychiatric Association)
* have any clinically important abnormality at screening, as determined by investigator, in physical or neurological examination, vital signs, electrocardiogram (ECG), or clinical laboratory test results that could be detrimental to the participant or could compromise the study.
* have a positive human immunodeficiency virus (HIV) test result at screening
* have a history of alcohol, illicit drug, analgesic or narcotic use disorder within 2 years prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Were Allocated to Each ISA | Baseline, Up to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (64):
- United States (62):
  - Central Research Associates, Birmingham, Alabama
  - Simon Williamson Clinic, Birmingham, Alabama
  - Synexus Clinical Research - Glendale, Glendale, Arizona
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - Irvine Clinical Research, Irvine, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - CMR of Greater New Haven, Hamden, Connecticut
  - VIN-Julie Schwartzbard, Aventura, Florida
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - K2 MEDICAL Research THE VILLAGES, Lady Lake, Florida
  - K2 Medical Research ORLANDO, Maitland, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - Flourish Research - Miami, LLC, Miami, Florida
  - University of Miami Don Suffer Clinical Research Building, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Synexus Clinical Research US, Inc., Orlando, Florida
  - Synexus Clinical Research - St. Petersburg, Pinellas Park, Florida
  - Martin E. Hale M.D., P.A., Plantation, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Synexus Clinical Research US, Inc., The Villages, Florida
  - Conquest Research, Winter Park, Florida
  - North Georgia Clinical Research, Woodstock, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Synexus Clinical Research, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Cotton O'Neil Clinical Research Center - Central Office, Topeka, Kansas
  - DelRicht Research, New Orleans, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Synexus Clinical Research US, Inc., Omaha, Nebraska
  - Rochester Clinical Research, LLC, Rochester, New York
  - PharmQuest, Greensboro, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Synexus - Cincinnati, Cincinnati, Ohio
  - Aventiv Research Inc, Columbus, Ohio
  - META Medical Research Institute, Dayton, Ohio
  - DelRicht Research, Tulsa, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading,LLC, Wyomissing, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - Synexus, Dallas, Texas
  - Cedar Health Research, Dallas, Texas
  - Re:Cognition Health - Fort Worth, Fort Worth, Texas
  - Synexus Clinical Research US, Inc., San Antonio, Texas
  - SYNEXUS, Murray, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Puerto Rico (2):
  - Ponce Medical School Foundation Inc., Ponce
  - Latin Clinical Trial Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Knopp KL, Downing AM, Anthony L, Chaterjee S, Price K, Sparks J. An innovative phase 2 chronic pain master protocol design to assess novel mechanisms in multiple pain types. Pain Rep. 2024 Oct 16;9(6):e1203. doi: 10.1097/PR9.0000000000001203. eCollection 2024 Dec. PMID 39430683

DOCUMENTS (1):
  • Study Protocol (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT05986292/Prot_005.pdf